CLINICAL TRIAL: NCT03415217
Title: Neighbourhood Team Development (NTD) Program
Acronym: NTD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Conestoga College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 137020
Record Dates: First submitted 2017-07-27; First posted 2018-01-30 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Nursing Homes; Quality of Health Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neighbourhood Team Development (Other): Neighbourhood Team Development consisted of a 30-month standardised training and implementation plan to promote inter-professional team collaboration and enhanced resident centeredness.
  Interventions: Other: Neighbourhood Team Development Program

INTERVENTIONS:
Other: Neighbourhood Team Development Program — The Neighbourhood Team Development Program aims to both enhance team development and resident centredness in LTC. The Program has three components, designed to modify the physical environment, the organization and delivery of services, and the alignment of staff members, to function independently and collaboratively in providing resident-centred care.

SUMMARY:
The purpose of this study is to evaluate the implementation and the effects of the Neighbourhood Team Development (NTD) Program, an innovative multi-component program that aims to provide resident centred care in long term facilities (LTC). As Canadians age, there is an increasing demand for LTC services. Older people residing in LTC homes and their families expect excellent care and services. However, literature and anecdotal evidence clearly indicate that LTC is not necessarily resident and family centred, nor are the care providers always collaborating as a team, thereby compromising the residents' quality of life.1-5 Residents with Alzheimer's Disease or Related Dementias (ADRD), who may have difficulty voicing their concerns, are at particular risk of receiving poor resident centred care.6,7 Decisions such as mealtimes in large dining rooms or early bedtimes are seldom in line with the residents' needs or wishes and add to the growing concern that the current LTC system is ill-designed and outdated. The NTD Program, designed by the investigators, aims to both enhance team development and resident centredness in LTC. The Program has three components, designed to modify the physical environment, the organization and delivery of services, and the alignment of staff members, to function independently and collaboratively in providing resident-centred care.

ELIGIBILITY:
* Long-stay resident, family member, or staff member in Schlegel Villages (chain of long-term care homes in Ontario, Canada)
* Able to obtain informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-05-15 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
The change in resident centredness (as assessed by the CARE Profile score) from baseline to 4 years | 4 years
  Linear regression adjusted for possible confounders including clustering of units in long-term care homes and case mix index.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Boscart VM, Sidani S, Ploeg J, Dupuis SL, Heckman G, Kim JL, d'Avernas J, Brown P. Neighbourhood Team Development to promote resident centred approaches in nursing homes: a protocol for a multi component intervention. BMC Health Serv Res. 2019 Dec 2;19(1):922. doi: 10.1186/s12913-019-4747-0. PMID 31791338